CLINICAL TRIAL: NCT05858047
Title: A Randomized, Double-blind, Placebo-controlled Phase Ⅱ Study to Evaluate the Efficacy and Safety of SYHX1901 Tablets in the Treatment of Moderate to Severe Plaque Psoriasis
Brief Title: An Investigational Study to Evaluate Experimental Medication SYHX1901 Tablets With Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYHX1902-002
Record Dates: First submitted 2023-03-03; First posted 2023-05-15 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Effects, Drug Side
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group I (Placebo) (Placebo Comparator): Placebo will be administered orally (PO) for 12 weeks.
  Interventions: Drug: Placebo
- Group Ⅱ (SYHX1901 60 mg) (Experimental): SYHX1901 will be administered orally (PO) for 12 weeks.
  Interventions: Drug: SYHX1901
- Group III (SYHX1901 90 mg) (Experimental): SYHX1901 will be administered orally (PO) for 12 weeks.
  Interventions: Drug: SYHX1901
- Group Ⅳ (SYHX1901 180 mg) (Experimental): SYHX1901 will be administered orally (PO) for 12 weeks.
  Interventions: Drug: SYHX1901

INTERVENTIONS:
Drug: Placebo — Administered orally, once daily (QD)
  Arms: Group I (Placebo)
Drug: SYHX1901 — Administered orally, once daily (QD)
  Arms: Group III (SYHX1901 90 mg); Group Ⅱ (SYHX1901 60 mg); Group Ⅳ (SYHX1901 180 mg)

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of different doses of SYHX1901 tablets in the treatment of moderate to severe plaque psoriasis in order to select doses for further clinical trials.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled phase Ⅱ study to evaluate the efficacy and safety of three different doses of SYHX1901 tablets compared with placebo in the treatment of moderate to severe plaque psoriasis. The total duration of the study will be 20 weeks which will be comprised of: a screening period (4 weeks); an efficacy assessment period (12 weeks) and a follow-up assessment period (4 weeks). Eligible subjects will be randomly assigned to SYHX1901 60 mg qd, 90 mg qd, 180 mg qd or placebo group at a 1:1:1:1 ratio for continuous oral administration for 12 weeks. The presence or absence of treatment with biological agents will be a stratification factor. Subjects will be monitored for the safety throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects fully understand and voluntarily participate in this study and sign informed consent;
2. Age ≥18 and ≤ 75 years old;
3. Subjects with a clinical diagnosis of stable moderate-to-severe plaque psoriasis with a history ≥6 months before randomization; Subjects with stable moderate-to-severe plaque psoriasis defined as meeting all four of the following criteria simultaneously:

   1. Subject must be diagnosed of chronic plaque psoriasis with no morphological changes or significant outbreaks of disease activity assessed by the investigator;
   2. Subject must be a candidate for systemic treatment or phototherapy assessed by the investigator;
   3. Body Surface Area (BSA) affected by plaque-type psoriasis ≥10% at screening and baseline;
   4. PASI score of ≥12 and Physician's Global Assessment (PGA) score ≥3 at screening and baseline;
4. Negative blood pregnancy results should be provided 14 days (inclusive) and 3 days (inclusive) prior to initial dosing, and subjects and their partners should voluntarily take contraceptive measures considered effective by the investigator during the study period and for at least 28 days after the study;
5. Subjects must be volunteer and be able to complete study procedures and follow-up examinations.

Exclusion Criteria:

1. Forms of psoriasis other than plaque psoriasis (Guttate psoriasis、erythrodermic psoriasis、Pustular psoriasis、Drug-induced psoriasis);
2. Previous or current autoimmune disease;
3. Other active skin conditions that may affect the clinical evaluation of psoriasis;
4. Active infection or fever at randomization;
5. Severe bacterial, fungal, or viral infection requiring hospitalization/intravenous drug treatment within 60 days prior to randomization;
6. Any proven history of untreated bacterial infection within 60 days prior to randomization;
7. Any existing evidence of chronic infection;
8. Any proven history of infection of a joint prosthesis or receiving antibiotics for a suspected joint prosthesis infection;
9. Received live vaccine within 60 days before randomization or scheduled to receive live vaccine within 60 days after the end of the study;
10. History of severe herpes zoster or sever herpes simplex infection;
11. Abnormal hepatitis B virus (HBV) related check during screening;
12. Hepatitis C virus (HCV) antibody positive at screening;
13. HIV antibody or treponema pallidum antibody positive;
14. Any known or suspected condition of congenital or acquired immunodeficiency;
15. Tuberculosis (TB);
16. Symptoms or signs of progressive or uncontrolled kidney, liver, blood, gastrointestinal, endocrine, lung, heart, neurological, psychiatric, or brain disease, or with other chronic diseases that the investigator has determined are not suitable for participation in this clinical trial;
17. History of malignancy or lymphoproliferative disease within 5 years (except for cured basal cell carcinoma and in situ cervical cancer);
18. Major surgery within 8 weeks before randomization or surgery planned during the study;
19. Uncontrolled hypertension, systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg after systemic treatment;
20. Having unstable cardiovascular disease defined as presence of a clinical cardiovascular event in the last 3 months or hospitalized for heart disease within the last 3 months; or NYHA≥3 grade, or abnormal ECG suggesting clinically significant and assessed by the investigator as carrying unforeseen risks;
21. History of arterial or venous thrombosis or at high risk;
22. Significant gastrointestinal disorders, such as erosion, hemorrhagic gastroenteritis, a history of bleeding from gastrointestinal ulcers, inflammatory bowel disease, and other disorders that investigator consider to be at risk for gastrointestinal perforation or that may interfere with drug ingestion, transport, or absorption;
23. Uncontrolled hyperlipidemia (TG>2.3 mmol/L and/or LDL>3.4 mmol/L) after standard treatment;
24. Low body weight (weight ≤45 kg or BMI≤18 kg/m^2);
25. BMI ≥30kg/m^2， (severe obesity);
26. Have received local anti-psoriasis therapy within 2 weeks prior to randomization; If topical moisturizers have been used within 2 weeks, they should be continued throughout the trial, with the same frequency and dose until the end of the study;
27. Have used physical therapy within 4 weeks prior to randomization (including photochemotherapy, ultraviolet therapy);
28. Systemic treatments:

    1. Systemic anti-psoriasis therapy within 4 weeks before study drug initiation;
    2. Leflunomide within 6 months before study drug initiation;
    3. Opioid analgesics within 4 weeks before study drug initiation;
    4. Lithium and antimalarial drugs within 4 weeks before study drug initiation;
    5. Any CYP3A4 potent inhibitor/inducer within 4 weeks before study drug initiation;
    6. Any P-gp potent inhibitor/inducer within 4 weeks before study drug initiation;
    7. Thymosin administered by injection or orally within 4 weeks before study drug initiation;
    8. Use of BCRP-sensitive substrate drugs assessed by the investigator during the study;
29. Biological agents:

    1. Exposure to any biological drug directly targeting IL-17 or IL-12, or IL-23 within 6 months prior to randomization ;
    2. Exposure to any TNF monoclonal antibody within 2 months prior to randomization;
    3. Exposure to any monoclonal antibodies against CD20 within 6 months prior to randomization;
    4. Exposure to any T cell or B cell modulators or integrin pathway modulators within 3 months prior to randomization;
    5. Any other biological drugs within 5 half-lives before study drug initiation;
30. Enrolled in a clinical study of any other drug within 3 months or use of any other investigational drugs within 5 half-lives of the investigational treatment before randomization;
31. History of lack of response to treatment after at least 3 months of treatment with any monoclonal antibody targeting IL-17 or IL-23 at approved doses;
32. Organ transplantation (except corneal transplantation more than 3 months before the initiation of the investigational drug);
33. Impossible to avoid prolonged daylight exposure during the trial, or to plan to use UV health rooms or other UV light sources;
34. Laboratory abnormalities of clinical significance assessed by the investigator to pose a risk:

    1. AST or ALT ≥ 2×ULN;
    2. Total bilirubin and/or direct bilirubin >2×ULN;
    3. Neutrophil absolute value (NEUT#) <1.5×10^9/L;
    4. Electrolyte imbalance;
35. History of alcohol and drug abuse or test positive for drug abuse;
36. History of neurological or psychiatric disorders, such as depression, suicidal tendencies, epilepsy, dementia, etc;
37. Any other medical and/or social reasons identified by the investigator as inappropriate for participation in the study;
38. Members of the research team and their immediate families.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2023-04-11 (Actual); Primary Completion 2024-02-21 (Actual); Study Completion 2024-02-21 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Achieving a Psoriasis Area and Severity Index Score ≥75% (PASI 75) response | Week 12

SECONDARY OUTCOMES:
Percentage of Participants Achieving a Psoriasis Area and Severity Index Score ≥50% (PASI 50) response | Week 12
Percentage of Participants Achieving a Physician Global Assessment (PGA) of 0 or 1 | Week 12
Change from Baseline in Body Surface Area (BSA) affected with Psoriasis to Week 12 | Week 12
Percentage of Participants Achieving a Dermatology Life Quality Index (DLQI) of 0 or 1 | Week 12

OTHER OUTCOMES:
Incidence of AEs and SAEs | Time Frame:Week 16

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No